CLINICAL TRIAL: NCT03411395
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Study to Evaluate the Efficacy of Different Doses of Amino Acids in 5AA+CrPic Water on Glucose Homeostasis in a Healthy Population.
Brief Title: Efficacy of Different Doses of Amino Acids in 5AA+CrPic Water on Glucose Homeostasis in a Healthy Population.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DoubleGood AB (Industry)
Collaborators: Lund University (Other); Aventure AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DG1603Lund
Record Dates: First submitted 2018-01-09; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: Diabetes; Prediabetes; Blood sugar regulation
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo drink (Placebo Comparator): A standardized breakfast meal will be provided together with carbonated water containing aroma
  Interventions: Other: Placebo drink
- 5AA+CrPic Water Dose 1 (Experimental): A standardized breakfast meal will be provided together with carbonated water containing aroma and active components 5AA and CrPic
  Interventions: Dietary Supplement: 5AA+CrPic Water
- 5AA+CrPic Water Dose 2 (Experimental): A standardized breakfast meal will be provided together with carbonated water containing aroma and active components 5AA (1/2 of Dose 1) and CrPic
  Interventions: Dietary Supplement: 5AA+CrPic Water
- 5AA+CrPic Water Dose 3 (Experimental): A standardized breakfast meal will be provided together with carbonated water containing aroma and active components 5AA (1/4 of Dose 1) and CrPic
  Interventions: Dietary Supplement: 5AA+CrPic Water

INTERVENTIONS:
Dietary Supplement: 5AA+CrPic Water — Dietary supplement drink with carbonation, aroma, amino acids and chromium picolinate
  Other Names: Good Idea
  Arms: 5AA+CrPic Water Dose 1; 5AA+CrPic Water Dose 2; 5AA+CrPic Water Dose 3
Other: Placebo drink — Placebo water with carbonation and aroma
  Arms: Placebo drink

SUMMARY:
It has previously been shown that a carbonated water including a defined amount of amino acids and chromium can decrease the postprandial glucose response. In this study, the effect of three different doses of amino acids on glucose excursions after a standardized test meal will be evaluated in healthy subjects. The study will be conducted in a randomized, single center, crossover, double-blinded, placebo controlled design including 25 participants. The primary endpoint of the study is the incremental area under the curve for capillary blood glucose (iAUC) within 180 minutes after ingestion of the meal.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18-25 (±0.5) kg/m²
* Agree to maintain consistent dietary habits and physical activity levels for the duration of the study
* Healthy as determined by medical history and information provided by the volunteer
* Willingness to complete questionnaires and follow instructions associated with the study and to complete all visits
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Pregnancy or lactation
* Known Type I or Type II diabetes
* Undetected Type I or Type II diabetes (fasting blood glucose < 6.1 mmol/L at first test day)
* Use of antibiotics
* Metabolic diseases and/or chronic gastrointestinal diseases (IBS, Crohns etc.)
* Allergy to test product or placebo ingredients
* Participants restricted to a vegetarian or vegan diet
* Intolerance to lactose or gluten
* Acute infection
* Individuals who are averse to venous catheterization or capillary blood sampling
* Alcohol or drug abuse
* Currently active smokers (tobacco products, and e-cigarettes)
* Participation in other clinical research trials
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the PI's opinion may adversely affect the individual's ability to complete the study or its measures or which may pose significant risk to the individual
* Any medical condition(s) or medication(s) known to significantly affect glucose metabolism. Significance to be assessed by the PI
* Use of medication, over-the-counter medication, natural health products or dietary supplements/probiotics that may affect glucose metabolism is prohibited during this study. Significance to be assessed by the PI. Participants who are taking allowed prescribed medications must agree to maintain their current method and dosing regimen during the course of the study unless recommended by their physician.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Blood glucose response | 3h postprandial phase
  The difference in three-hour incremental area under the curve (AUC) for capillary blood glucose between 5AA+CrPic test products and placebo following a standardized breakfast meal.

SECONDARY OUTCOMES:
Cmax of capillary blood glucose | 3h postprandial phase
  The difference in the three-hour Cmax (0 - 180 min) of capillary blood glucose between 5AA+CrPic test products and the placebo following a standardized meal.
Serum insulin response | 3h postprandial phase
  The difference of the three-hour iAUC (0 - 180 min) intravenous serum insulin iAUC between 5AA+CrPic test products and the placebo following a standardized meal.
Venous blood glucose response | 3h postprandial phase
  The difference of the three-hour iAUC (0 - 180 min) intravenous plasma glucose iAUC between 5AA+CrPic test products and the placebo following a standardized meal.
GLP-1 response | 1h postprandial phase
  The difference of the 1h iAUC (0 - 60 min) intravenous blood glucagon-like peptide 1 (GLP-1) iAUC between 5AA+CrPic test products and the placebo following a standardized meal.
Capillary blood glucose response | 2h postprandial phase
  The difference in the two-hour iAUC (0 - 120 min) capillary blood glucose iAUC between 5AA+CrPic test products and the placebo following a standardized meal.

CONTACTS AND LOCATIONS:
Overall Officials: Elin Östman, PhD, Principal Investigator — Scheelevägen 22 223 63 Lund, Sweden; Kristina Andersson, PhD, Study Director — Experimental Medical Science, Lund University, Sweden; Lovisa Heyman-Lindén, PhD, Study Chair — Scheelevägen 22 223 63 Lund, Sweden